CLINICAL TRIAL: NCT06323122
Title: A Comparative Study Between Three Different Plating Techniques in Management of Mandibular Parasymphyseal Fractures. A Retrospective Study
Brief Title: A Comparative Study Between Three Different Plating Techniques in Management of Mandibular Parasymphyseal Fractures.
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Nermine Ramadan Mahmoud, Associated Professor of oral and maxillofacial surgery, Oral Surgery Department, October 6 University
Other Study IDs: Plating Techniques 2023
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Mandibular Fractures
Keywords: parasymphyseal; mandibular fracture; internal fixation; miniplates; 3D miniplate
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group (I): ORIF was done using two 2.0 miniplates
  Interventions: Device: 2.0 miniplates
- Group II: ORIF was done using 2.3 high profile miniplates
  Interventions: Device: 2.3 high profile miniplates
- Group III: ORIF was done using 3D miniplates.
  Interventions: Device: 3D miniplates

INTERVENTIONS:
Device: 2.0 miniplates — 2.0 miniplates
  Groups: group (I)
Device: 2.3 high profile miniplates — 2.3 high profile miniplates
  Groups: Group II
Device: 3D miniplates — 3D miniplates
  Groups: Group III

SUMMARY:
The main goal in management of mandibular fractures is to restore the pre-injury form and function, with the least disability and shortest recovery period.

DETAILED DESCRIPTION:
Currently there are a diversity of metallic hardware used for fixation of jaw fractures. However, the proper selection of the suitable technique is still a matter of debate.

The aim of the current study was to compare between the effect of two miniplates, 2.3 high profile Miniplates and three dimensional (3D) Miniplates for internal fixation treatment of mandibular para-symphyseal fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symphyseal/ parasymphyseal mandibular fracture.
2. Patients presenting within 7 days of trauma.

Exclusion Criteria:

1. Associated fractures that could affect occlusion or dimensions
2. Medically compromised patients who are unfit for management under General Anesthesia
3. Patients with gross infection at the site of fracture
4. Patients not willing to return for follow-up
5. Patients with associated bone pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who had suffered from a recent mandibular fractures in the symphyseal or parasymphyseal region which required Open Reduction with Internal Fixation (ORIF)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Surgery Time | intraoperative
  measure the time of surgery from incision till closure with minutes

SECONDARY OUTCOMES:
complication | 6 months
  record the surgical complication operative and postoperative
fracture stability | 6 months
  measure fracture stability from radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Nermine Ramadan Mahmoud, PhD, Principal Investigator — Associated Professor of oral and maxillofacial surgery, Oral Surgery Department
Locations (1):
- October 6U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu W, Agrawal M, Thadani S, Mukul SK, Sood R, Patel A, Dhanak R, Tailor S. Comparative evaluation of a single 2.0-mm AO locking reconstruction plate with conventional miniplate osteosynthesis for treatment of linear non-comminuted fractures of symphysis and parasymphsis region of the mandible. J Stomatol Oral Maxillofac Surg. 2019 Feb;120(1):11-15. doi: 10.1016/j.jormas.2018.10.002. Epub 2018 Oct 26. PMID 30739640